CLINICAL TRIAL: NCT00296413
Title: Variation of Serum Valproate and Lamotrigine Levels in Relation to The Menstrual Cycle and Oral Contraceptive Use
Brief Title: A Study to Look at Antiepileptic Drug Levels While on Lamictal or Depakote With or Without an Oral Contraceptive
Status: Completed | Type: Observational
Sponsor: Beth Israel Deaconess Medical Center (Other)
Collaborators: Rhode Island Hospital (Other)
Responsible Party: Principal Investigator, Andrew Herzog, Professor of Neurology, Beth Israel Deaconess Medical Center
Other Study IDs: 2005P000379
Record Dates: First submitted 2006-02-21; First posted 2006-02-27 (Estimated); Last update posted 2017-03-14 (Actual); Status verified 2017-03

CONDITIONS: Epilepsy
Keywords: epilepsy; menstrual cycle; valproate; lamotrigine; oral contraceptive
MeSH Terms: conditions — Epilepsy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Serum Samples for hormone testing
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (4):
- 1: Valproate monotherapy
- 2: Valproate monotherapy with combined oral contraceptive
- 3: Lamotrigine monotherapy
- 4: Lamotrigine monotherapy with combined oral contraceptive

SUMMARY:
Some antiseizure medication levels are affected by hormones. This study is being done to determine if blood levels of lamotrigine or valproate are affected by the hormones in the birth control pill or the menstrual cycle itself.

DETAILED DESCRIPTION:
Participants will be given informed consent and will be asked to have two blood draws at specific times of the menstrual cycle or if on a birth control pill, during the active and inactive pill phases.

ELIGIBILITY:
Inclusion Criteria:

* Must be a female between 13-45 years of age
* Must have a history of seizures
* Must be taking either lamotrigine (Lamictal) or valproate (Depakote) with or without a birth control pill

Exclusion Criteria:

* Must not be on antidepressant medication, tranquilizers, or other forms of hormonal therapy other than the birth control pill

Ages: 13 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Two regional epilepsy centers
Sampling Method: Non-Probability Sample
Enrollment: 48 (Estimated)
Dates: Start 2006-02; Primary Completion 2009-02 (Actual); Study Completion 2009-02 (Actual)

PRIMARY OUTCOMES:
To carry out a controlled investigation to determine if combined oral contraceptive (COC) use affects serum valproate (VPA) and lamotrigine (LTG) levels | 3 years
To distinguish any apparent COC effects from the potential effects of the naturally occurring high (mid luteal) and low (early follicular, menstrual) steroid phases of the menstrual cycle itself | 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Andrew G. Herzog, M.D., M.Sc., Principal Investigator — Beth Israel Deaconess Medical Center
Locations (1):
- Beth Israel Deaconess Medical Center, Boston, Massachusetts, United States